CLINICAL TRIAL: NCT00811551
Title: zWedge Clinical Feasibility IDE Study
Brief Title: Data Collection Study of Wedge Pressure Data in Patients With CRT-D Devices
Acronym: zWedge
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD 440
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Impedance Monitoring; Wedge Pressure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CRT-D (Intra-thoracic Impedance Monitoring) — Diagnostic Feature in CRT-D device that emits a sub-threshold pulse to measure resistance between two electrodes.

SUMMARY:
zWedge is a clinical feasibility IDE study. The objective is to characterize the relationship between intra-thoracic impedance measurements obtained from a CRT-D device and pulmonary capillary wedge pressure (PCWP) measured via a right heart catheterization (RHC) acutely and over time.

DETAILED DESCRIPTION:
Intra-thoracic impedance will be obtained at programmed intervals by using an investigational monitoring feature in the CRT-D device. To obtain impedance values, the device delivers a sub-threshold impulse that measures the resistance between 2 electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Have a SJM PROMOTE CRT-D (Model 3207 or other model with similar functioning) system that was implanted at least 4 months prior to enrollment for an approved indication per ACC/AHA/HRS guidelines.
* Have the ability to provide written informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluation.
* Have legally marketed bipolar right atrial and true bipolar right ventricular pacing defibrillation leads, and a legally marketed endocardial bipolar LV lead.

Exclusion Criteria:

* Be less than 18 years of age.
* Have any medical condition that would interfere with intra-thoracic measurements such as end-stage pulmonary disease, advanced interstitial pulmonary disease, or frequent episodes of pneumonia.
* Have a contraindication for right heart catheterization.
* Have a contraindication for the delivery of IV Nitroglycerin.
* Be pregnant or planning a pregnancy for the duration of their study participation.
* Be currently participating in a clinical investigation that includes an active treatment arm.
* Have a life expectancy of less than 12 months due to any condition.
* Be unable to perform the Valsalva maneuver with airway pressure > 40 mm Hg for ≥10 seconds.
* Are pacemaker dependent, where cessation of pacemaker function consistently results in syncope or ventricular asystole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously implanted with a St. Jude Medical PROMOTE device (Model 3207 or other with similar capability) according to ACC/AHA/HRS guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Carlson, MD, Study Director — Abbott Medical Devices
Locations (7):
- United States (7):
  - Little Rock Cardiology Clinic, Little Rock, Arkansas
  - Huntington Memorial Hospital, Pasadena, California
  - Colorado Springs Cardiology, Colorado Springs, Colorado
  - The Emory Clinic - Crawford Long Hospital, Atlanta, Georgia
  - Midwest Heart Research Foundation, Lombard, Illinois
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - St. Thomas Hospital Heart, Nashville, Tennessee